CLINICAL TRIAL: NCT03332953
Title: Sensory Perception of Sweet Flavors in E-Cigarette
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Responsible Party: Principal Investigator, Juyun Lim, Associate Professor, Oregon State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB # 8252
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Electronic Nicotine Delivery Systems; Flavoring Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- E-cigarette (Other): Subjects will be asked to vape various e-cigarettes at three concentrations of nicotine and sweet flavor (9 stimuli per subject). The subject will be asked to make ratings for the overall liking or disliking of the e-cigarette, followed by ratings on perceived intensities of sensations.
  Interventions: Other: E-cigarettes with varying concentrations of nicotine & flavor

INTERVENTIONS:
Other: E-cigarettes with varying concentrations of nicotine & flavor — Subjects will be asked to vape various e-cigarettes containing e-liquids at three concentrations of nicotine and sweet flavor (9 stimuli per subject).

SUMMARY:
Despite the explosive popularity of sweet flavored electronic cigarettes, there is little empirical evidence regarding how "sweet" flavors interact with different levels of nicotine to reduce its perceived bitterness and harshness, and thereby increase its appeal and additive potential. This study will serve to fill this knowledge gap through empirical psychophysical data that will determine the association between sweet flavor and nicotine and its link to the acceptance and rejection of vaped nicotine.

DETAILED DESCRIPTION:
We will recruit current, healthy e-cigarette users between the ages of 18-35.This study will require 1 visit to the Oregon State University campus to partake in a 1 hour (approximate) testing session. During the testing session, participants will be asked to puff commercial e-cigarettes containing 9 commercially available e-liquid preparations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18-35 years of age; have been vaping for at least 1 month; currently use an e-cigarette that contains nicotine; have used an e-cigarette with medium (9-12 mg/mL) or high (18 to 36 mg/mL) nicotine strength at some point in their e-cigarette using history.

Exclusion Criteria:

* Do not have mouth or throat problems that would keep subject from vaping comfortably; do not have health problems that would keep subject from tasting or smelling normally; do not have any food ingredient allergies and have never had an allergic reaction to propylene glycol or vegetable glycerin; do not have any respiratory allergies (i.e., frequent sneezing, nasal congestion, nasal discharge); do not have a history of pulmonary disease or asthma; are not in the process of trying to quit vaping; are not pregnant, breast feeding, or trying to become pregnant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Hedonic and Intensity Ratings | Until July 2018
  The outcome will be ratings obtained for liking or disliking of the stimulus and ratings for perceived intensities of sensations. These quantitative values collected from the scaling procedure will be analyzed corresponding to the level of nicotine and flavor for the particular stimulus. For rating perceived intensity, we will use the general Labeled Magnitude Scale (gLMS), developed for measurement of the intensity of oral sensation and taste. The scale is bounded by 'no sensation' at the bottom to 'strongest imaginable sensation of any kind' on top, with intermediate ratings between (bottom to top: barely detectable, weak, moderate, strong, very strong). A Labeled Hedonic Scale (LHS) will be used to measure individuals' liking or disliking of the oral sensation. The scale encompasses from "most disliked sensation imaginable" on one end to "most liked sensation imaginable" on the other end, with intermediate hedonic labels (like/dislike: slightly, moderately, very much, extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Juyun Lim, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT03332953/ICF_000.pdf